CLINICAL TRIAL: NCT00481299
Title: Insulin Resistance and Lipid Profile in Non-Obese Women With Prolactinoma Treated With Dopamine Agonists
Brief Title: Insulin Resistance in Women With Prolactinoma
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Other Study IDs: 178/04
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-04

CONDITIONS: Prolactinoma; Insulin Resistance; Hyperlipidemia
Keywords: Insulin; glucose; lipids; prolactinoma; hyperprolactinemia
MeSH Terms: conditions — Prolactinoma; Insulin Resistance; Hyperlipidemias; Hyperprolactinemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prolactin is suggested to influence insulin resistance, but scarce data is available on the metabolic profile of patients with prolactinoma.

The purpose of the protocol was to evaluate cardiovascular disease risk factors in women with prolactinoma treated with dopamine agonists and to study the influence of disease control and anthropometry on their metabolic profile.

DETAILED DESCRIPTION:
A cross-sectional study was performed in non-obese premenopausal women with prolactinoma treated with dopamine agonists evaluated regarding glucose, insulin, Homeostasis Model Assessment (HOMA), lipid profile, C reactive protein (CRP), body mass index (BMI), waist circumference, prolactin, estradiol, testosterone, and sex hormone binding globulin (SHBG). They were compared with control women of similar age and BMI distribution.

ELIGIBILITY:
Inclusion Criteria:

* Prolactinoma
* Female gender
* Premenopausal

Exclusion Criteria:

* Obesity (BMI ≥ 30 kg/m²)
* Diabetes mellitus
* Hypertension
* GH deficiency
* Hypothyroidism
* Primary hypogonadism
* Adrenal insufficiency
* Pituitary surgery

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2004 (Actual)
Dates: Start 2004-10; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika CO Naliato, MSc, Principal Investigator — Federal University of Rio de Janeiro - Brazil
Locations (1):
- Clementino Fraga Filho University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil